CLINICAL TRIAL: NCT00487890
Title: Performance Evaluation and Research for Older Adults Requiring Major Surgery
Acronym: PERFORM
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Flum, Professor, Surgery, University of Washington
Other Study IDs: 25699
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Geriatric; Abdominal; Surgery; gastrointestinal surgery; intrabdominal surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to identify modifiable factors in older adults associated with functional decline following major non-emergent surgery. The hypothesis of this proposal is that poor preoperative exercise tolerance and physical performance, potentially modifiable factors, are crucial in predicting functional decline and disability following surgery. When completed, this study will reveal detailed information on the incidence and risk factors for functional decline in older adults following surgery. It will direct future research targeting interventions in older adults at highest risk for functional decline following surgery, thereby decreasing the incidence of premature disability.

DETAILED DESCRIPTION:
This prospective cohort study will follow 400 patients undergoing major non-emergent abdominal or cardiothoracic surgery at the University of Washington Medical Center. Patients 65 and older will be recruited following introduction of the study by a health-care provider. The provider will give the patient a study pamphlet and letter outlining the study. Patients who express interest in the study will meet with a Research Coordinator. The Coordinator will describe the study, answer all questions, and have the patient review and provide written informed consent. The Mini-cog, a validated brief dementia screen with high sensitivity and specificity, will be used to determine if patients have a potential cognitive impairment. Participants who recall all 3 words correctly or draw a normal clock will be considered cognitively intact and able to provide consent and to participate in the study. Participants who are unable to recall any words or who draw an abnormal clock will be ineligible for the study and classified as having a potential cognitive impairment.

Consenting patients will be asked questions about their medical history and health status. The Research Coordinator will only ask questions that are relevant to the patient's medical care. The 5-item version of the Geriatric Depression Scale will assess patients for active depression. This short version has been validated and found to be highly sensitive and specific for diagnosing depression. Patients will also be asked to complete the Duke Activity Status Index and the Health Assessment Questionnaire. These questions will take 10-15 minutes.

Patients will be asked to perform physical tasks. These tasks will include a physical performance measure. Patients will only be asked to complete tasks that they are comfortable performing. The physical performance measures include 1) a timed 10-ft walk at normal pace, 2) a timed test of repetitive chair stands, 3) a hierarchial balance task, and 4) testing of grip strength. In the timed walk, patients are asked to walk at normal pace for 10 feet. This task is completed twice with the average of the times calculated. In the timed test of 5 repetitive chair stands, patients are asked to fold their arms across their chest and to rise from the seated position 5 times as quickly as possible. To assess balance, patients are asked to stand with their feet side-by-side, followed by semi-tandem, and tandem and to hold each position for 10 seconds. Scores are allotted based upon how far each participant is able to progress. To test grip strength, a handheld dynamometer will be used. Using an isometric dynamometer, the best score of the 3 squeezes from the dominant hand will be the value calculated.

Patients will be asked to complete the EQ-5D, SF-36 and Health Assessment Questionnaires at 1 week, 1 month, 3 months and 12 months following their surgery as well as the CNAQ Appetite Questionnaire but only at the 1 month, 3 month, and 1 year follow up intervals. The Research Coordinator will contact them by phone to complete these questionnaires. If the patient is still in the hospital at the University of Washington 1 week following their surgery, the Research Coordinator will meet with them to complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older;
* Having abdominal surgery;
* Informed consent obtained;
* All races/ethnicities;
* Both genders

Exclusion Criteria:

* Non-English speaking;
* Unwillingness to participate;
* Unavailable for follow-up phone calls;
* Unable to communicate with researchers;
* Unable to pass the screening test

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults, aged 65 and older, who are undergoing an abdominal or cardiothoracic surgical procedure at the University of Washington Medical Center in Seattle, WA.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States